CLINICAL TRIAL: NCT07377201
Title: How Do Adults With Cerebral Palsy Perceive Their Botulinum Toxin Treatment During Childhood ?
Brief Title: Childhood Toxin Perception Survey
Acronym: PERTOXE
Status: Recruiting | Type: Observational
Sponsor: Centre Médico-Chirurgical de Réadaptation des Massues Croix Rouge Française (Other)
Responsible Party: Sponsor
Other Study IDs: 2025_09_PERTOXE_RIPH3; 2025-A01186-43 (Other: ID-RCB)
Record Dates: First submitted 2025-12-29; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy (CP)
MeSH Terms: conditions — Cerebral Palsy | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with cerebral pasly previously treated with botulinum toxin
  Interventions: Other: Patient-Reported Outcome Measures

INTERVENTIONS:
Other: Patient-Reported Outcome Measures — Participants will complete questionnaires regarding their perception of childhood botulinum toxin injections and their current coping strategies. No new medical treatment is administered.

SUMMARY:
Context:

Most medical and surgical interventions for individuals with Cerebral Palsy (CP)-such as botulinum toxin injections, orthopedic surgery, and rehabilitation-occur during childhood. While these treatments are costly and resource-intensive, there is a significant lack of long-term data regarding their effectiveness in adulthood. Furthermore, the perspective of adult patients on the care they received as children is rarely documented. Understanding this "patient-centered" perspective is vital, as care aligned with an individual's values is proven to result in higher satisfaction and better health outcomes.

Problem Statement While botulinum toxin (BTX) has been the gold standard for treating focal spasticity since 2009, it is an iterative (repeated) treatment that can involve procedure-induced pain. At present, there is limited knowledge about how adults with CP perceive the long-term impact of childhood vaccinations. The emotional and physical burden of repeated treatments during development is also not well understood, as are the coping strategies developed by these individuals to manage the stress and pain associated with long-term medical care.

Objectives

The PERTOXE study is a prospective study designed to explore the transition from childhood care to adult life for individuals with CP. Its primary goals are:

Perception of Care: To evaluate how adults with CP perceive the effectiveness and impact of the botulinum toxin injections they received during childhood.

Lived Experience: To document the subjective experience of treatment, including induced pain and the quality of communication with healthcare providers.

Coping Mechanisms: To explore the "coping strategies" these individuals use to face stressful medical events and chronic functional decline.

Significance As the lifespan of individuals with CP increases, understanding long-term outcomes is a research priority. By collecting data from adults, this study aims to improve current pediatric practices, ensuring that childhood interventions better support a high quality of life, functional maintenance, and psychological well-being in adulthood.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years or older
* Diagnosed with cerebral palsy
* Received repeated toxin injections during childhood (> 2 series of injections)
* Agreeing to complete the questionnaire
* Possessing sufficient cognitive abilities, particularly in terms of reading comprehension and oral comprehension (even if someone had to physically assist them in responding)
* All levels of the GMFCS classification 1 to 5

Exclusion Criteria:

* Individuals who do not meet the above criteria, as confirmed by the statements in Part 1 of the survey, will be automatically excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with cerebral palsy who experienced botulinum treatment during childhood
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Treatment experience | At enrollment
  This assessment is not based on a single scale, but on a series of multidimensional questions exploring the patient's memories on the treatment they received in childhood:
  * Induced pain: Assessment of the pain relief methods used (MEOPA, EMLA, anaesthesia, etc.).
  * Communication and preparation: Questions about the quality of preparation, how well the medical team listened, the consent process, and understanding of the purpose of the treatment.
  * Overall satisfaction: Use of satisfaction scales from 0 to 10 (where 0 = 'not at all satisfied' and 10 = 'perfectly satisfied') to rate effectiveness, conditions and communication.

SECONDARY OUTCOMES:
Coping Strategies BRIEF-Cope Scale | At enrollment
  Use of the French version of the BRIEF-Cope (28 items) to identify the specific coping mechanisms (e.g., active coping, denial, humor, or substance use) used by adults with Cerebral Palsy when facing stressful events.
  Respondents use a 4-point scale to answer each statement: 1 - not at all; 2 - a little; 3 - a lot; 4 - very much.
  The responses obtained are added up for each scale. Higher scores on a scale indicate increased use of that coping mechanism.

CONTACTS AND LOCATIONS:
Locations (1):
- CMCR des Massues, Lyon, France